CLINICAL TRIAL: NCT02760030
Title: Phase II Trial of Primary Endocrine Therapy With Combination of Fulvestrant or an Aromatase Inhibitor and Palbociclib in Elderly Patients With Hormone Responsive Breast Cancer Who Have Inoperable Tumor Or Operable Tumor But Cannot Undergo Surgery Due to Frailty Or Who Refuse Surgery
Brief Title: Endocrine Therapy Fulvestrant & Palbociclib or Aromatase Inhibitor Therapy in Treating Older Patients With Hormone Responsive Breast Cancer That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Nicole Williams, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-15266; NCI-2016-00146 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2016-03-29; First posted 2016-05-03 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-10

CONDITIONS: Estrogen Receptor and/or Progesterone Receptor Positive; HER2/Neu Negative; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; palbociclib; Aromatase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (fulvestrant, palbociclib) (Experimental): Patients receive fulvestrant IM on days 1 and 15. Patients also receive palbociclib PO QD on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Fulvestrant; Other: Laboratory Biomarker Analysis; Drug: Palbociclib; Other: Questionnaire Administration; Drug: Aromatase Inhibitors

INTERVENTIONS:
Drug: Fulvestrant — Given IM
  Other Names: Faslodex; Faslodex(ICI 182,780); ICI 182,780; ICI 182780; ZD9238
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Palbociclib — Given PO
  Other Names: Ibrance; PD-0332991; PD-332991
Other: Questionnaire Administration — Correlative studies
Drug: Aromatase Inhibitors — Given PO

SUMMARY:
This phase II clinical trial studies how well fulvestrant and palbociclib works in treating older patients with breast cancer that responds to hormone treatment (hormone responsive) that cannot be removed by surgery. Estrogen can cause the growth of estrogen-receptor-positive breast cancer cells. Hormone therapy using fulvestrant may fight estrogen-receptor-positive breast cancer by blocking the use of estrogen by the tumor cells. Palbociclib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving fulvestrant together with palbociclib may be an effective treatment for hormone responsive breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine treatment failure-free survival (TFFS) rate at one year of combination therapy with pure estrogen antagonist, fulvestrant and cyclin-dependent kinase (CDK) inhibitor, palbociclib as primary endocrine therapy in patients 70 years or older with newly diagnosed non-metastatic hormone receptor positive, human epidermal growth factor receptor 2 (HER-2) negative breast cancer.

SECONDARY OBJECTIVES:

I. To determine 1- and 2-year progression free survival. II. To determine safety and toxicity of this combination in the population of patients 70 years or older.

III. To determine whether longitudinal changes in geriatric assessment measures correlate with tolerability of this regimen.

OUTLINE:

Patients receive fulvestrant intramuscularly (IM) on days 1 and 15. Patients also receive palbociclib orally (PO) once daily (QD) on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed invasive, estrogen receptor (ER) and/or progesterone receptor (PR)-positive, HER2 negative breast cancer; ER-and/or PR-positive breast cancer is defined by > 10% staining by immunohistochemistry
* Patients must be vulnerable or frail by Balducci Criteria or the patient is refusing breast surgery; vulnerable patients are defined as those with dependence in some instrumental activities of daily living, well controlled co-morbidities, and early symptoms of geriatric syndrome; frail patients are defined as those with three or more co-morbidities, dependence in one or more activities of daily living, or a clinically significant geriatric syndrome; geriatric syndromes include: dementia, delirium, incontinence (fecal and/or urinary), osteoporosis or spontaneous fractures, polypharmacy, visual/hearing impairment, sarcopenia and neglect or abuse
* The patient's refusal to proceed with curative breast surgery has to be documented by the surgeon's and medical oncologist's note
* Absolute neutrophil count (ANC) > 1000/uL
* Platelets > 75,000/L
* Serum creatinine 1.5 X institutional upper limit of normal (ULN)
* Total bilirubin < 1.5 X ULN
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) 2.5 ULN
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior aromatase inhibitor therapy
* Evidence of distant metastases
* Psychiatric illness, which would prevent the patient from giving informed consent
* Patients receiving strong inducers or inhibitors of cytochrome P450 3A4 (CYP3A4)

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Treatment failure-free survival (TFFS) defined as the proportion of study subjects who remain on treatment from the 1st day of therapy to one year | 1 year
  The proportion of subjects who do not experience treatment failure at one year will be calculated along with the exact binomial confidence interval for the rate.

SECONDARY OUTCOMES:
Change in cognition, as measured by Blessed Orientation-Memory-Concentration Test | Baseline to up to 12 weeks after removal from study
  Comprehensive geriatric assessment measures to assess functional independence will be summarized using descriptive statistics such as proportions with confidence intervals and means with standard deviations.
Change in comorbidities, as measured by the Charlson comorbidity index | Baseline to up to 12 weeks after removal from study
  Comprehensive geriatric assessment measures to assess functional independence will be summarized using descriptive statistics such as proportions with confidence intervals and means with standard deviations.
Change in depression, as measured by the Geriatric Depression Scale | Baseline to up to 12 weeks after removal from study
  Comprehensive geriatric assessment measures to assess functional independence will be summarized using descriptive statistics such as proportions with confidence intervals and means with standard deviations.
Change in functional status, as measured by the ECOG Performance Status Scale | Baseline to up to 12 weeks after removal from study
  Comprehensive geriatric assessment measures to assess functional independence will be summarized using descriptive statistics such as proportions with confidence intervals and means with standard deviations.
Change in functional status, as measured by the History of falls | Baseline to up to 12 weeks after removal from study
  Comprehensive geriatric assessment measures to assess functional independence will be summarized using descriptive statistics such as proportions with confidence intervals and means with standard deviations.
Change in functional status, as measured by the Timed Up test | Baseline to up to 12 weeks after removal from study
  Comprehensive geriatric assessment measures to assess functional independence will be summarized using descriptive statistics such as proportions with confidence intervals and means with standard deviations.
Change in functional status, as measured by the Go Test | Baseline to up to 12 weeks after removal from study
  Comprehensive geriatric assessment measures to assess functional independence will be summarized using descriptive statistics such as proportions with confidence intervals and means with standard deviations.
Change in functional status, as measured by the Instrumental Activities of Daily Living | Baseline to up to 12 weeks after removal from study
  Comprehensive geriatric assessment measures to assess functional independence will be summarized using descriptive statistics such as proportions with confidence intervals and means with standard deviations.
Change in nutritional status, as measured by the Mini Nutritional Assessment | Baseline to up to 12 weeks after removal from study
  Comprehensive geriatric assessment measures to assess functional independence will be summarized using descriptive statistics such as proportions with confidence intervals and means with standard deviations.
Change in social activity and support, as measured by the Medical Outcome Study (MOS) | Baseline to up to 12 weeks after removal from study
  Comprehensive geriatric assessment measures to assess functional independence will be summarized using descriptive statistics such as proportions with confidence intervals and means with standard deviations.
Change in social activity and support, as measured by Social Activity Limitations Survey. | Baseline to up to 12 weeks after removal from study
  Comprehensive geriatric assessment measures to assess functional independence will be summarized using descriptive statistics such as proportions with confidence intervals and means with standard deviations.
Incidence of adverse events, using the National Cancer Institute Common Terminology Criteria for Adverse Events version 4 | Up to 12 weeks after removal from study
  The proportion of adverse events and the exact binomial confidence interval for the rates will also be calculated.
Progression free survival | Up to 1 year
  Calculated using Kaplan-Meier methods.
Progression free survival (PFS) | Up to 2 years
  Calculated using Kaplan-Meier methods

CONTACTS AND LOCATIONS:
Overall Officials: Nicole O Williams, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (3):
- United States (3):
  - St. Elizabeth Healthcare, Edgewood, Kentucky
  - Case Western University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu